CLINICAL TRIAL: NCT04523584
Title: Ultrasound Quantification of Liver Fat
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: CIN_US Liver Fat
Record Dates: First submitted 2020-08-14; First posted 2020-08-21 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-06

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Magnetic Resonance Imaging; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Hepatic Steatosis: <5% liver fat fraction by MRI PDFF
  Interventions: Device: Magnetic Resonance Imaging (MRI); Device: Ultrasound Imaging
- No Hepatic Steatosis: >5% liver fat fraction by MRI PDFF
  Interventions: Device: Magnetic Resonance Imaging (MRI); Device: Ultrasound Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging (MRI) — Participants will undergo MR imaging of the liver. Liver PDFF will be measured.
Device: Ultrasound Imaging — Participants will undergo ultrasound imaging of the liver. UDFF and shear wave speed (US-SWS) will be measured.

SUMMARY:
The investigators plan a prospective study designed to evaluate the accuracy of a new ultrasound method for quantification of liver fat content.

DETAILED DESCRIPTION:
MRI proton density fat fraction (PDFF) will serve as the reference standard for liver fat fraction measurements. The strength of agreement between ultrasound derived fat fraction (UDFF) and PDFF will be the outcome of interest for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients 16 years of age or older with known fatty liver disease (based upon prior MRI or ultrasound), or at risk for fatty liver disease (obese).

Exclusion Criteria:

* Subject under the age of 16
* Pregnant subject
* Subjects who cannot cooperate with performance of the ultrasound exam
* Subjects who cannot cooperate with performance of the MRI exam
* Subjects who have contraindications to MRI
* Subjects who might require sedation or anesthesia to undergo study imaging

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients 16 years of age or older with known fatty liver disease (based upon prior MRI or ultrasound), or at risk for fatty liver disease (obese).
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
MRI PDFF correlation/agreement to UDFF | Single time point-30 minute MRI/30 minute Ultrasound
  Liver fat % derived using MR PDFF will be compared to UDFF

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanquinet S, Rougemont AL, Courvoisier D, Rubbia-Brandt L, McLin V, Tempia M, Anooshiravani M. Acoustic radiation force impulse (ARFI) elastography for the noninvasive diagnosis of liver fibrosis in children. Pediatr Radiol. 2013 Mar;43(5):545-51. doi: 10.1007/s00247-012-2595-8. Epub 2012 Dec 28. PMID 23271404
- [Background] Fierbinteanu Braticevici C, Sporea I, Panaitescu E, Tribus L. Value of acoustic radiation force impulse imaging elastography for non-invasive evaluation of patients with nonalcoholic fatty liver disease. Ultrasound Med Biol. 2013 Nov;39(11):1942-50. doi: 10.1016/j.ultrasmedbio.2013.04.019. Epub 2013 Aug 9. PMID 23932277
- [Background] Kinner S, Reeder SB, Yokoo T. Quantitative Imaging Biomarkers of NAFLD. Dig Dis Sci. 2016 May;61(5):1337-47. doi: 10.1007/s10620-016-4037-1. Epub 2016 Feb 5. PMID 26848588
- [Background] Middleton MS, Van Natta ML, Heba ER, Alazraki A, Trout AT, Masand P, Brunt EM, Kleiner DE, Doo E, Tonascia J, Lavine JE, Shen W, Hamilton G, Schwimmer JB, Sirlin CB; NASH Clinical Research Network. Diagnostic accuracy of magnetic resonance imaging hepatic proton density fat fraction in pediatric nonalcoholic fatty liver disease. Hepatology. 2018 Mar;67(3):858-872. doi: 10.1002/hep.29596. Epub 2018 Jan 26. PMID 29028128
- [Background] Trout AT, Dillman JR, Xanthakos S, Kohli R, Sprague G, Serai S, Mahley AD, Podberesky DJ. Prospective Assessment of Correlation between US Acoustic Radiation Force Impulse and MR Elastography in a Pediatric Population: Dispersion of US Shear-Wave Speed Measurement Matters. Radiology. 2016 Nov;281(2):544-552. doi: 10.1148/radiol.2016152797. Epub 2016 May 26. PMID 27228332
- [Background] Tyagi A, Yeganeh O, Levin Y, Hooker JC, Hamilton GC, Wolfson T, Gamst A, Zand AK, Heba E, Loomba R, Schwimmer J, Middleton MS, Sirlin CB. Intra- and inter-examination repeatability of magnetic resonance spectroscopy, magnitude-based MRI, and complex-based MRI for estimation of hepatic proton density fat fraction in overweight and obese children and adults. Abdom Imaging. 2015 Oct;40(8):3070-7. doi: 10.1007/s00261-015-0542-5. PMID 26350282
- [Derived] Dillman JR, Thapaliya S, Tkach JA, Trout AT. Quantification of Hepatic Steatosis by Ultrasound: Prospective Comparison With MRI Proton Density Fat Fraction as Reference Standard. AJR Am J Roentgenol. 2022 Nov;219(5):784-791. doi: 10.2214/AJR.22.27878. Epub 2022 Jun 8. PMID 35674351